CLINICAL TRIAL: NCT03455790
Title: An Investigation of the Relationship Between Upper Extremity Muscle Strength, Anaerobic Capacity, Aerobic Capacity and Sportive Performance in Wheelchair Basketball Athletes
Brief Title: Relationship Between Muscle Strength,Anaerobic,Aerobic Capacity,and Sportive Performance in WC Basketball Athletes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 640
Record Dates: First submitted 2018-02-27; First posted 2018-03-07 (Actual); Last update posted 2018-03-07 (Actual); Status verified 2018-03

CONDITIONS: Sports Physical Therapy
Keywords: Wheelchair Basketball,; Isokinetic; Anaerobic Capacity; Shoulder Muscle Strength; Aerobic Capacity,; Sportive Performance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Wheelchair Basketball (Experimental): Upper limb muscle strength assessments of the athletes will be performed with the ISOMED 2000® isokinetic device and the grip strength with the Jamar® dynamometer. The aerobic capacity values will be measured using the Cosmed K5® instrument and the TS in the Cosmos-Saturn brand running band. Anaerobic capacity will be measured by Wingate anaerobic power test (WanT) for 30 seconds in standard laboratory conditions for TS basketball athletes using Monark 894 E model ergometer developed by Monark for upper extremity anaerobic capacity and power measurement. The sporty performances will be evaluated with the "20 m Sprint test", "Slalom Test" and "Zone Shot" tests.
  Interventions: Diagnostic Test: Aerobic Capacity
- 20 Meters Sprint Test (Experimental): It will be done to evaluate the speed of sportsmen's wheelchair use. The sportsman will be prompted to take the chair as fast as possible after the wheelchair has been positioned so that the front bar is on the field edge. The 2 meter slow-down distance will also be counted in seconds and the completion time of the 20 meter track will be measured.
  Interventions: Diagnostic Test: Aerobic Capacity
- Slalom test (Other): It will be done to measure the ability of sportsmen to use wheelchairs. Five cones will be placed starting 1.5 meters from the starting line of the Sahara, with a distance of 1.5 meters between them. Sportsmen will be required to complete the course by making a slalom between these topics and making a slalom in the same way by turning back and passing through the starting line. Track completion times will be recorded in seconds.
  Interventions: Diagnostic Test: Aerobic Capacity
- Zone Shot Test (Other): Zone Shot test will be applied to evaluate the shooting skills of the athletes. In the starting position the athlete will be asked to shoot the pot from the athlete with the warning given while on the foul shooting line and then to take their own rebounds. They will have to shoot again from the point where they have taken the rebound and rebound and go back to the foul line. The test will continue for 2 minutes in this manner. At the end of the 2-minute training period, the athletes will score the correct shot 2, the missed shot 1 point and the total score will be recorded.
  Interventions: Diagnostic Test: Aerobic Capacity
- Aerobic Capacity (Other): To measure aerobic capacity values, it shall be measured with Cosmed K5® device and Cosmos-Saturn branded treadmill using TS which is used in routine workout with customized ramp protocol. Before starting the test, the athlete's TS walking belt at a speed of 1 mph (1.7 km / h) at 0% incline for 3 min. and it will be checked whether or not the gas measuring equipment is disturbing the participant. If the athlete is unable to continue, the time at which the test will end will be determined. Time min. . The air that the individual exposes during the test will be collected using a breath by breath method.
  Interventions: Diagnostic Test: Aerobic Capacity
- Anaerobic Capacity (Other): Using the Monark 894 E model ergometer developed by Monark for upper extremity anaerobic capacity and power measurement, TS basketball athletes will be subjected to a Wingate anaerobic power test (WanT) for 30 seconds in standard laboratory conditions.
  Interventions: Diagnostic Test: Aerobic Capacity
- Isokinetic shoulder muscle strength (Other): Upper limb muscle strength assessments of the athletes will be performed with the ISOMED 2000® isokinetic device and the grip strength with the Jamar® dynamometer.
  Interventions: Diagnostic Test: Aerobic Capacity

INTERVENTIONS:
Diagnostic Test: Aerobic Capacity — Upper limb muscle strength assessments of the athletes will be performed with the ISOMED 2000® isokinetic device and the grip strength with the Jamar® dynamometer. The aerobic capacity values will be measured using the Cosmed K5® instrument and the TS in the Cosmos-Saturn brand running band. Anaerobic capacity will be measured by Wingate anaerobic power test (WanT) for 30 seconds in standard laboratory conditions for TS basketball athletes using Monark 894 E model ergometer developed by Monark for upper extremity anaerobic capacity and power measurement. The sporty performances will be evaluated with the "20 m Sprint test", "Slalom Test" and "Zone Shot" tests.
  Other Names: Anaerobic Capacity; Sportive Performance; Zone Shot Test; Slalom Test; 20 Meters Sprint Test

SUMMARY:
The aim of the study is to investigate the relationship between shoulder internal and external rotation isokinetic muscle strength, grip strength, anaerobic capacity, aerobic capacity and sportive performance in wheelchair basketball athletes. Through this work, we aim to contribute to the literature with objective, blood-based results.

The wheelchair (WC) basketball characterizes high intensity activities such as rolling, rebounding, rolling, smashing overhead. Because these activities are fast and powerful, they require both anaerobic and aerobic capacities. The main factors affecting WC Basketball performance are upper extremity muscle strength and aerobic capacity. It is stated that higher muscle power and aerobic performance in WC Basketball will provide more independence in daily life activities as well as increased speed and power during sports play.

WC basketball players have both a spore-specific activities and a shoulder rotational muscle strength aerobic power components have a critical functional role when using a wheelchair. When the literature on this subject is examined, it is seen that there is a limited number of works for WC basketball sport which is very popular nowadays. Assessment of upper limb muscle strength, aerobic capacity and sporting performance in wheelchair basketball athletes is crucial in regulating the athletes' training programs and establishing individual training programs.

DETAILED DESCRIPTION:
This study was aimed to investigate the relationship between isokinetic muscle strength of shoulder internal and external rotation, grip strength, anaerobic capacity, aerobic capacity and sportive performance in wheelchair basketball athletes.

26 wheelchair basketball athletes were involved into the study. Wheelchair basketball players were divided into two groups according to the classification levels (Group 1: less than 3 points, Group 2: 3 points and higher). Upper extremity muscle strengths were evaluated with the ISOMED 2000® isokinetic device. Hand grip strength was evaluated with hydraulic hand dynamometer. The measurement of the aerobic capacity was measured using its own wheelchair on the treadmill by applying a custom ramp protocol. Anaerobic capacity was evaluated with Wingate anaerobic power test (WAnT) for 30 seconds in standard laboratory conditions. The sportive performances were assessed by "20 m Sprint test", "Slalom Test" and "Zone Shot" tests.

ELIGIBILITY:
Inclusion Criteria:

* Professional and / or competitor measurement athlete playing TS basketball for at least one year

  * Being between the ages of 18-45
  * Approving participation in written work as self-employed or legal representative
  * Possibility of co-oping the parameters to be applied in the study
  * There is no health problem between their own

Exclusion Criteria:

* • Have undergone surgery with upper extremity and / or upper body in the past 6 months

  * Acute shoulder pain
  * Leaving the sport for at least 3 months, not actively participating in the training
  * Partial or complete finger loss in the upper extremity, congenital deformity and contractures, spasticity
  * Having a previously identified and diagnosed condition (cardiovascular, etc.)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 26 (Actual)
Dates: Start 2017-11-25 (Actual); Primary Completion 2017-12-30 (Actual); Study Completion 2018-01-18 (Actual)

PRIMARY OUTCOMES:
Evaluation of Isokinetic Muscle Strength | 1 months
  0-90 ° scapular planda concentric-concentric with 10 repeats of 60 ° / sec in the direction of IR and ER. fast and 15 repetitions 180 ° / sec. maximal shoulder internal and external rotation movements were done bilaterally

CONTACTS AND LOCATIONS:
Overall Officials: ÇAĞLAR SOYLU, postgraduate, Principal Investigator — Ankara Yıldırım Beyazıt University, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation
Locations (1):
- Ankara Yıldırım Beyazıt University, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation, Ankara, Etlik, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No